CLINICAL TRIAL: NCT02068248
Title: Effect of Viscous Soluble Fibers on Serum Cholesterol Levels: A Series of Systematic Reviews and Meta-analyses
Brief Title: Effect of Viscous Soluble Fibers on Serum Cholesterol Levels
Acronym: CHOL-META
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: Cholesterol Meta
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: LDL Cholesterol

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: Soluble Fibre

SUMMARY:
Research over the past several decades have linked the intake of dietary fiber with lower blood cholesterol levels. The distinction between soluble and insoluble fiber fractions emerged shortly after and there is now a general consensus that soluble fiber possesses the capacity to lower cholesterol. Since the discovery of the cholesterol lowering effects of soluble dietary fiber, there has been much debate as to the degree of cholesterol reduction from these fibers. In order to handle the inconsistencies a full and systematic review of the published literature was conducted by Brown et. al (1999). Results from this meta-analysis, concluded that 'increasing soluble fiber can make only a small contribution to lowering cholesterol.'

Research is constantly progressing and new research findings may not always be consistent with older data. For example, results from new research are now challenging the previously approved health claims for soy foods and fatty acids. This is a major public health concern because if clinical evidence is not reliable, it could lead to harm. Since the publication of the meta-analysis by Brown et. al (1999) over a decade ago, scientists have continued to research the effects of soluble fiber on cholesterol levels with new technology and trial designs, therefore it is crucial to revisit the question and update the literature on the effect of viscous soluble dietary fibers on serum cholesterol levels.

A series of meta-analyses will be performed to assess the link between viscous dietary fibers and serum cholesterol levels. Nutritionists now consider fiber to be an integral part of diet and disease. Results from these meta-analyses help address the question of whether viscous soluble fibers have a role lowering serum cholesterol levels.

ELIGIBILITY:
Inclusion Criteria:

* Randomized Controlled Trials
* Paralell or Crossover Design
* Duration: >3 weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: No Restrictions
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Serum LDL Cholesterol Level | 3 weeks

SECONDARY OUTCOMES:
Serum Non-HDL Cholesterol Level | 3 weeks
Serum Apolipoprotein B Level | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Unity Health Toronto; John Sievenpiper, MD, PhD, Principal Investigator — Unity Health Toronto; Thanh Ho, MSc (C), Study Director — Unity Health Toronto
Locations (1):
- The Toronto 3D Knowledge Synthesis and Clinical Trials Unit, Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Ho HVT, Jovanovski E, Zurbau A, Blanco Mejia S, Sievenpiper JL, Au-Yeung F, Jenkins AL, Duvnjak L, Leiter L, Vuksan V. A systematic review and meta-analysis of randomized controlled trials of the effect of konjac glucomannan, a viscous soluble fiber, on LDL cholesterol and the new lipid targets non-HDL cholesterol and apolipoprotein B. Am J Clin Nutr. 2017 May;105(5):1239-1247. doi: 10.3945/ajcn.116.142158. Epub 2017 Mar 29. PMID 28356275